CLINICAL TRIAL: NCT04315350
Title: The Effect of Curcumin on the Development of Prednisolone-induced Hepatic Insulin Resistance in Overweight and Obese Participants
Brief Title: The Effect of Curcumin on the Development of Prednisolone-induced Hepatic Insulin Resistance
Acronym: CURPRED
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We stopped recruiting having 8 in each intervention group instead of 9 due to recruitment problems due to COVID19 pandemic
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Pernille Høgh Hellmann, Medical Doctor, primary investigator, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-19017550
Record Dates: First submitted 2020-01-14; First posted 2020-03-19 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Insulin Resistance; Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Insulin Resistance; Non-alcoholic Fatty Liver Disease | interventions — Prednisolone

STUDY DESIGN:
Intervention Model Description: After study day 1, participants are randomized (1:1:1) to one of three treatments: 1) Prednisolon and Curcumin, 2) Prednisolon and placebo or 3) Placebo and placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Curcumin (Experimental): Participant receives both curcumin and prednisolone. Curcumin for 11 days, prednisolone for 10 days. Curcumin: 2 tablets (each contains 100 mg curcumin) twice daily. Prednisolon: 50 mg (capsule) every morning
  Interventions: Drug: Curcumin Liposome
- Prednisolon (Other): Participant receives prednisolone and curcumin-placebo. Curcumin-placebo for 11 days, prednisolone for 10 days. Curcumin-placebo: 2 tablets twice daily. Prednisolon: 50 mg (capsule) every morning
  Interventions: Drug: Prednisolone
- Placebo (Placebo Comparator): Participant receives prednisolone.placebo and curcumin-placebo. Curcumin-placebo for 11 days, prednisolone-placebo for 10 days. Curcumin-placebo: 2 tablets twice daily. Prednisolon-placebo: One capsule every morning.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Curcumin Liposome — Curcumin is given together with prednisolone
  Arms: Curcumin
Drug: Prednisolone — Prednisolone is given together with curcumin-placebo
  Arms: Prednisolon
Drug: Placebos — Prednisolone-placebo is given together with curcumin-placebo
  Arms: Placebo

SUMMARY:
The aim of this study is to investigate whether ingestion of curcumin will prevent hepatic insulin resistance (assessed by homeostatic model assessment of insulin resistance (HOMA-IR)) induced by short-term oral glucocorticoid (prednisolone) administration in overweight and obese participants. As a secondary endpoint it will be investigated if prednisolone administration induce or worsen the degree of NAFLD in overweight or obese participants using magnetic resonance (MR) spectroscopy (MRS), and if curcumin can ameliorate this effect. Also, the possible anti-inflammatory effect of curcumin will be elucidated as a range of inflammatory markers before and after intervention will be measured. Thus, prednisolone treatment is used as a model of development of pre-diabetes.

DETAILED DESCRIPTION:
AIMS OF STUDY The aim of this study is to investigate whether ingestion of curcumin will prevent hepatic insulin resistance (assessed by homeostatic model assessment of insulin resistance (HOMA-IR)) induced by short-term oral glucocorticoid (prednisolone) administration in overweight and obese participants.

BACKGROUND The increasing incidence and prevalence of obesity and its comorbidities calls for research in preventing these diseases. The progression to insulin resistance and increased blood sugar levels (i.e. prediabetes) and ultimately type 2 diabetes (T2D) in obesity is believed to be caused by various factors of which low-grade inflammation in adipose tissue and skeletal muscle tissue seems to inflict insulin resistance initiating metabolic deterioration towards the type 2 diabetic phenotype. Curcumin, a polyphenolic compound that can be extracted from the turmeric root, have been shown to exert anti-inflammatory properties in both in vitro and animal studies. Furthermore, animal studies indicate that curcumin is a modulator of gut microbiota composition in a metabolic beneficial direction. Studies have shown positive results in terms of lowering hepatic insulin resistance with curcumin in rodents and humans (measured by HOMA-IR), and another clinical trial has shown that curcumin can prevent worsening of HOMA-IR and development of T2D in a prediabetic population.

Glucocorticoids are a group of frequently used compounds, prescribed for a wide range of diseases and have severe metabolic side effects as insulin resistance, T2D and non-alcoholic fatty liver disease. Interestingly, curcumin, a phenolic compound extracted from the turmeric root, and curcumin analogues have been shown to ameliorate glucocorticoid-induced 'dysmetabolism' in rodent studies, but no human data exist. Also, results from both in vitro and in vivo studies with curcumin have shown promising effects in preventing NAFLD development, but solid human data are missing. Because of the temporary effects on glucose metabolism, short-term treatment with glucocorticoids can be used as an investigative model of these metabolic changes. Previous studies from the research unit performing the current study, used this setup to investigate changes in glucose homeostasis, incretin hormones and insulin resistance. Two different mouse studies indicate that curcumin could be beneficial in terms of preventing the metabolic changes associated with systemic glucocorticoid treatment, but no human studies have investigated if curcumin can prevent glucocorticoid-induced increase in HOMA-IR.

The aim of the study is to investigate the effects of curcumin of the metabolic changes caused by short-term systemic prednisolone in a double-blinded, placebo-controlled trial in overweight and obese individuals.

STUDY DESIGN

Participants 27 overweight and obese individuals without diabetes

METHODS

In this randomised, double-blinded, placebo-controlled trial, eligible participants will undergo baseline assessments before being randomised to one of the following interventions: 1) Two tablets of curcumin (each tablet containing 100 mg curcumin) twice daily in 11 days and 50 mg of prednisolone once daily in 10 days (capsule); 2) two tablets of placebo-curcumin twice daily in 11 days and 50 mg of prednisolone once daily in 10 days (capsule); 3) two tablets of placebo-curcumin twice daily in 11 days and one capsule of placebo-prednisolone once daily in 10 days. In the end of the 11-day intervention period, end-of-intervention assessments (similar to baseline assessments) will be performed. If necessary, a follow-up visit will be made.

Information meeting and screening Prior to any protocol-related procedures, an information meeting will be arranged, and participants will be informed of the possibility of bringing a person of own choice to the visit. The information meeting is performed in undisturbed and confidential surroundings. The room is reserved for this purpose, and nobody will interfere during the meeting. It is not possible for other employees in the department to look into the room. During this meeting, a member of the research group will explain the purpose, procedures and possible risks of the study. The member of the research group will have proper qualifications in terms of medical knowledge, insights in the specific project and communications skills. It is firstly pointed out that the project is a biomedical trial. After this, an oral information about the project is given based on the written information. Questions will be answered as thoroughly as possible. The participant will be informed that it is possible to have a minimum of 48 hours to evaluate participation from oral information is given. If he does not want time to evaluate the participation, the informed consent can be obtained. If he wants time to evaluate participation, a new meeting will be arranged with a minimum of 48 hours from the information meeting. When the informed consent has been obtained, screening can be done, either the same day or another day, but with a maximum of four weeks after obtaining the informed consent. The participant will be informed that it is possible to withdraw the written consent at any time prior to or during the study. In the case that significant information about the participants health is found during the trial, the participant will be able to decline having this information. Information about this choice is confirmed in the informed consent form.

If the participant wants to know about the results of the trial and the possible consequences for the participant, he will have the rights to get this information after the end of the study At screening, height and body weight will be measured, medication and medical history will be recorded, blood will be sampled for assessment of plasma/serum concentrations of thyroid-stimulating hormone, creatinine, creatine kinase, electrolytes, aspartate aminotransferase (ASAT), alanine aminotransferase (ALAT), lactate dehydrogenase, alkaline phosphatase, albumin, bilirubin, gamma-glutamyltransferase, viral hepatitis markers, platelet count, ferritin and haemoglobin, and albumin-creatinine ratio in the urine will be measured. A physical examination will be made including evaluation of blood pressure and pulse rate. Alcohol habits will be evaluated based on The Alcohol Use Disorder Identification Test (AUDIT) questionnaire and quantification of the weekly amount of alcohol. An MR safety checklist will be completed, and an MR information sheet will be given. If all inclusion criteria and none of the exclusion criteria are met, dates for baseline assessments and randomisation visit will be planned within 6 weeks from the screening visit. The participant will be instructed not to consume curcumin-containing food on a daily basis from screening until end of trial.

Baseline assessments and randomisation visit

If the participant is included during COVID19 pandemic, a phone call is done the day before the visit to ask about recent symptoms of infection, contacts to people with COVID19 symptoms or people with positive test for COVID19.

Included individuals will undergo an MRS of the liver (scheduled as close as possible to the randomisation visit). Before intervention start, both randomisation visit and MRS will be performed. For MRS, participants are placed in a horizontal position. During the MRS, a spectroscopy of the liver will be assessed, and an estimation of visceral adipose tissue and subcutaneous adipose tissue will be done.

During the last week before randomisation, the subject will collect a stool sample for the determination of gut bacteria count and subtype. Stool samples will be collected by the participant at home. Prior to defaecation a disposable collector will be placed in the toilet from where stool will be transferred to a tube that immediately is transferred to a transport container and placed at -20°C in the patient's freezer. Prior to transport to Gentofte Hospital, the transport container is transferred to the cooler bag and at arrival at Gentofte Hospital the transport container (with the sample tube) is immediately stored in at -80°C for later analysis. This entails DNA extraction, library preperation, MiSeq 16S rRNA sequencing and microbiota analysis (relative abundance, alpha/beta diversity, link to phenotype of interest).

On the randomisation visit, the participant will meet in the laboratory around 8 a.m. after 10 hours of fast (including any medication) and refrainment from tobacco or nicotine supplements use. The participant is allowed to drink water until 8 hours before meeting in department. Furthermore, the participant will be requested to avoid heavy alcohol intake (more than 5 units of alcohol per day) and strenuous exercise two days prior to the visit and instructed to use non-strenuous methods of transportation to the research facility. The following procedures will be conducted:

If the test day is during COVID19 pandemic, the participant is tested for Sars-Cov2 with a swab procedure in the oropharynx, for immidiate PCR analysis.

1. A fasting urine sample will be collected, and the participant is asked to empty the urinary bladder completely
2. Fasting blood samples will be collected (bone markers, serum markers of muscle breakdown, biomarkers of NASH and fibrosis, fibroblast growths factors, triglycerides, cholesterols, liver parameters, HbA1c, inflammatory markers, adipokines, creatinine, haemoglobin) amounting 25 ml.
3. FibroScan: The participant will be lying in a supine position for approximately 10 minutes during which a probe using shear-waves and ultrasound is applied in the right side of the body below the ribs.
4. Measurement of blood pressure, heart rate, body weight and hip and waist circumference.
5. A questionnaire is handed out regarding calorie intake and physical activity the day prior to randomisation
6. IOP is measured with icare ic100 tonometer.
7. One cannula will be inserted in the cubital vein for collection of blood samples. The forearm from which blood samples are drawn will be wrapped in a heating blanket (42°C) throughout the experiment (for arterialisation of venous blood).
8. Blood samples (for analysis of total amino acids, gut hormones, glucose, glucagon, insulin, C-peptide, urea, FFA) will be measured throughout the OGTT (see Table 1).
9. At time 0 min, the participant will ingest 75 g of water-free glucose dissolved in 300 ml water over a period of 5 minutes.
10. At time 0, 30, 60, 90, 120, 150, 180, 210, 240 and after the ad libitum meal, hunger, satiety, fullness and prospective food consumption will be measured by VASs
11. During the last hour (time 180 min - 240 min), REE will be measured in a supine position by indirect calorimetry to determine oxygen consumption (V02) and carbon dioxide production (VC02). A flow-through canopy gas analyser will be used, as previously described.
12. At time 240 min, the subject will be asked to provide a new urine sample for measurement of urea concentration. The participant will be asked to empty the urinary bladder completely. Urine volume will be measured.
13. At time ~250 min, the participant will ingest a standardised ad libitum meal consisting of minced meat, pasta, corn, carrots, peppers, cream, salt and pepper (50 energy (E)% carbohydrate, 37 E% fat, 13 E% protein). The participant will be instructed to eat as much as possible until feeling comfortable saturate. The meal should be consumed within a maximum of 30 minutes and by the end of the meal, time spent eating, weight of the meal and the total amount of energy consumed will be noted.
14. A continuous glucose monitor will be applied on the upper arm of the participant. The sensor is blinded which means that the participant cannot see his blood glucose excursions during the 14 days period of measurements.

At the end of the randomisation visit, the participant will be randomly assigned to one of three interventions (1:1:1):

1. Two tablets of curcumin (corresponding to 200 mg) twice daily from day 1 to day 11 and prednisolone capsule 50 mg (oral) once daily from day 2 to day 11
2. Two tablets of placebo-curcumin twice daily from day 1 to day 11 and prednisolone capsule 50 mg once daily from day 2 to day 11, or
3. Two tablets of placebo-curcumin twice daily from day 1 to day 11 and placebo-prednisolone capsule once daily from day 2 to day 11 The tablets with curcumin and placebo-curcumin will appear identical, and the capsules with prednisolone or placebo-prednisolone will appear identical.

The supplier of curcumin will also produce placebo-curcumin tablets (Indena Aps, Milan, Italy). The pharmacy of Region H will be responsible of production and delivery of prednisolone and placebo-prednisolon. Unblinded site-staff will be responsible for labelling and blinding of the curcumin and placebo-curcumin tablets and prednisolone and placebo-prednisolone capsules before the beginning of the intervention period. A person not otherwise involved in the study will generate a randomisation code using a random list generator. A randomisation list with randomisation numbers and corresponding treatment will be made by the unblinded site-staff. A list with randomisation number and corresponding packages with numbers will be made by unblinded site-staff, so that blinded site staff is only allocating a randomisation number at the day of randomisation. The list with the information about randomisation number and corresponding treatment will be kept at Center for Clinical Metabolic Research at Gentofte Hospital. If a participant develops adverse events (AEs) that demand knowledge of the content of the intervention, the list will show if the patient is having any active ingredients. If a participant is excluded of the trial before end-of-intervention visit, a new subject will be included in the same treatment-arm by taking over the randomisation number.

The interventional period If the participant was tested for Sars-Cov2-infection at randomization visit, this test has to be negative before start of intervention. If the participant is included during COVID19 pandemic, a telephone call is made the day before intervention start, to ensure the following guidelines are followed: If the participant has experiences symptoms of COVID19 during the last seven days prior to intervention start or had close contact with COVID19-patients, intervention will not be started.

Intervention will start soon after baseline MRS and randomisation visit. During the intervention period, each participant will fill out a dairy to keep track of any new concomitant medication, compliance and possible AEs. The participant will be asked to keep the alcohol and smoking habits they might have had before screening and, thus, not to consume more than 21 units of alcohol per week. Furthermore, they will be asked to consume no more than 5 units in one night. The participant will be requested to maintain the level of physical activity from before intervention during the interventional period. The participant will be informed that if he feels more hungry than usual, he is allowed to eat extra. At day 5, 6 or 7 in the intervention period, the participant will receive a telephone call from the investigator or other delegated site staff, checking on AEs, concomitant medication and compliance, and to answer any questions from the participant. Furthermore, participants are instructed to contact investigator or other delegated site staff in case of any questions or intolerable side effects.

The tablets and capsules are preferably ingested with a meal and a small glass of water. Should the participant forget to take a dose of curcumin/placebo curcumin, it can be ingested until 6 hours before the next planned dose. If a dosage is missed, and the next one is planned within 6 hours, the dosage should be passed, and the incident must be noted in the diary. Should the participant forget to take a dose of prednisolone/placebo-prednisolone, it can be ingested until 12 hours prior to the next dose. If a dosage is missed, and the next one is planned within the next 12 hours, the dosage should med passed, and the incident must be noted in the diary.

If the participant is included during COVID19 pandemic: The participant is instructed to adhere to social distancing and to be aware of COVID19-symptoms, and call site staff in any case of symptoms during intervention period or if he has had close contact to a person who had a positive Sars-Cov2-test, and to immediately stop intake of intervention and self-isolate in this case.

End-of-intervention assessments and visit The end-of-intervention visit will be planned on day 12 after start of intervention. If the participant is included during COVID19 pandemic, a telephone call is done the day before the visit to ask about recent symptoms of COVID19, recent contacts to people with COVID19 symptoms or people with positive test for COVID19.

Stool sample collection and MRS will be performed in the period around end-of-intervention visit, and will be performed as described above under "baseline assessments and randomisation visit". Procedures during the end-of-intervention visit are similar to the ones described above under "Baseline assessments and randomisation visit". Also, during this day, to check for any effect of curcumin intervention, physical examination will be performed by a physician from the research team and additional blood samples (identical with the samples at the screening visit, except viral hepatitis markers) will be collected (which adds another 5 ml blood samples compared to randomisation visit) and albumin-creatinine ratio in the urine will be measured. The continuous glucose monitor sensor is removed from the upper arm of the participant, and the data from the sensor is transferred to a suitable software program. Again, the questionnaire is handed out regarding calorie intake and physical activity the day prior to the End-of-intervention day. Compliance will be evaluated (if compliance is insufficient (missed more than ¼ of planned doses), the participant will not go through end-of-intervention assessments). If the participant is included during COVID19 pandemic, he is instructed to continue social distancing for three days after end-of-intervention visit.

Follow-up phone call and visit Between two and four days after last day on treatment, the participant will receive a telephone call, where the participant is asked about withdrawal symptoms and symptoms of COVID19. Due to COVID19, an extra telephone call is made at day 5-8 after end-of-intervention visit.

If the participant feels any kind of withdrawal symptoms (tiredness, weakness, abdominal pain, anorexia, nausea or vomiting), or has had any symptoms of an ongoing infection after End-of-intervention, a plan of action is made. Judged from the physical examination, blood tests, results from continuous glucose monitoring, MRS and FibroScan at End-of-intervention visit, a follow-up visit will be arranged, if it - judged by the investigator - is necessary. At this follow-up visit (3-4 weeks after End-of-intervention) the investigator can do any or all of the following tests; physical examination, FibroScan, measurement of IOC, standard OGTT and blood tests, whichever is judged to be necessary to look into any late effects of the intervention, and if necessary, another follow-up visit after another 1-3 months. If the participant had steatosis on both MRS's, the participant will be offered a referral to the Department of Gastroenterology for further evaluation and treatment.

BIOBANK A research biobank will be established at at Center for Clinical Metabolic Research at Gentofte Hospital, DK-2900 Hellerup, Denmark, during the experiments to store the blood tests until analyses. All participants are assigned with a trial number and will on data sheets and tubes only appear with the trial number. The full name, social security number and trial number will be stored separately. After the project is completed the biobank will be terminated. Excess plasma will be stored in another biobank for up to 10 years after the completion of the study, in case of need of re-analyses or need for further analyses. In the latter case, a new approval by the Regional Health Research Ethics Committee is required. The biobanks will be registered with Datatilsynet.

CALCULATIONS AND STATISTICS Data will be processed and presented with the use of standard descriptive statistics. Areas under the curves (AUCs) are calculated by use of the trapezoid rule. Comparison of normally distributed data is carried out by means of repeated measurements analysis of variance using linear mixed modeling with "individual" as random factor. Freidmans test will be used for analysis of non-normally distributed data. P values ≤0.05 are accepted as statistically significant (significance level, α = 5%). Power of the study (1-β) is set to 80%, where β (20%) is the risk of accepting a hypothesis that is false.

Power calculation: Hansen et al. studied a prednisolone-treated group of healthy individuals, and found an increase in HOMA-IR of 1.6 (1.3±0.1 vs. 2.9±0.3). The difference is 1.6±SD, but the value of this SD we unfortunately do not have. Best guess is that it is (maximum) 0.5. It is hypothesized that the intervention group receiving two different kinds of placebo is comparable to the baseline values in KB Hansens study, both before and after intervention, as placebo expectedly will not change HOMA-IR. And it is hypothesized that the prednisolone treated group is comparable with KB Hansens cohort after treatment with prednisolone. The wish is to achieve a reduction in the increase in HOMA-IR of 50% when ingesting curcumin, which gives a minimal relevant difference of 0.8.

P values ≤ 0.05 are accepted as statistically significant (α = 5%) and the power is set to 80%. This results in a sample size of 7 in each of the three treatment groups. . Based on this, we will include 9 in each of the three treatment groups, as we might have slightly more variance in HOMA-IR in our population compared to KH Hansen's participants. In case of drop-outs, we will include new participants until we have 12 completers in each group.

The continuous glucose monitoring will provide data for up to 14 days with glucose measures with frequent intervals 24 hours per day. The CGM will be recording for at least 24 hours before start of intervention with prednisolon. CGM recordings are regarded successful if at least 80% of the sensor data are available for analysis. Before analysis, all data will be reviewed for pressure induced sensor attenuations. From these data, the following calculations will be made: 1) The risk of hypoglycemia and hyperglycemia will be calculated as the low blood glucose index (LBGI) and the high blood glucose index (HBGI) using the EasyGV workbook (www.phc.ox.ac.uk/research/technology-outputs/easygv) 2) coefficient of variability (SD/mean interstitial glucose level), 3) SD, 4) percentage of time in normoglycemic range (3,9-7,8 mmol/l), 5) percentage of time in three hyperglycemic ranges (7.9-10 mmol/l, 10.1-13.9 mmol/l, >13.9mmol/l) and 6) percentage of time in hypoglycemia (<3.9 mmol/l).

SIDE EFFECTS, RISKS AND DISADVANTAGES FOR PARTICIPANTS Curcumin is a polyphenolic compound extracted from the turmeric root with a very low bioavailability. High doses of Meriva® have been well tolerated in human trials. However, most studies have been performed with non-formulated traditional curcumin with lower bioavailability. Nevertheless, high doses of non-formulated curcumin have not been associated with severe side effects, and are generally very well tolerated in clinical trials. Panahi et al did a study with NAFLD patients, with ~50 patients receiving Meriva® 1000 mg daily for 8 weeks (corresponding to 200 mg of curcumin). There were no reports of side effects, but 7 withdraw because of the perception of lack of effects. Antiga et. al. did a study with Meriva® 2000 mg daily for 12 weeks, with only one participant having one adverse event (diarrhoea), but presumably not caused by Meriva® because of other signs of viral genesis67. Mazzolani did a study with 12 patients receiving 1200 mg Meriva® per day for 1 year with no reports of AEs. Di Pierro et al. did a study on overweight participants, with a high dose of phosphatidylserine (a product very similar to Meriva®) with reports of no side effects.

Prednisolone side effects are very well described, and most commonly are weight gain, skin abnormalities, increased serum glucose levels, insulin resistance, oedema, electrolyte derangement, myopathy, osteoporosis, infections, reduced symptoms of infections, haematological abnormalities, psychiatric diseases, mood changes, sleep disorders, hyperlipidaemia, hypertension and heart failure. But if the participants will experience side effects, they are unlikely to get severe, when treating only with 50 mg daily for 10 days, as they are dose and time-dependent, and with the relevant inclusion and exclusion criteria applied. Furthermore, they are all regarded as fully reversible after end of intervention.

A side effect from treatment with oral corticosteroids (e.g. Prednisolone) is elevated IOP which in rare cases can cause the sight-threatening condition, glaucoma. In most cases elevated IOP is asymptomatic, which is why, it is important to measure in the patient. IOP can simply and easily be measured with a icare ic100 tonometer. The device is based on a rebound measuring principle that requires no drops, air or specialized skills for its use, and therefore not associated with any risk or complications. IOP is measured 3 times in each eye and the mean is calculated. If this is elevated the patient will be seen by an ophthalmologist.

During and right after prednisolone treatment, the participants are more prone to infections and are likely to have fewer symptoms of infections. Participants will be asked about their wellbeing and symptoms of infection several times during the trial.

If the participant is included during the COVID19 pandemic, several extra restrictions and assessments are applied in the study, due to the possible increased risk of a severe course of COVID19 in case of prednisolone treatment. This is applied only to take extraordinary precautions. Information on these restrictions and assessments is found in the relevant parts of this protocol. Participants are thoroughly instructed in the relevant changes in the participant information documents before screening.

Withdrawal symptoms (after prednisolone treatment) are most commonly tiredness, weakness, abdominal pain, anorexia, nausea or vomiting. Due to the short treatment period and relatively low dose, it is very unlikely these symptoms will occur, but participants will be asked about these symptoms at the telephone call two to four days after last day on treatment.

MRS is safe and not coupled with discomfort or pain. The scanner will be making loud noise while scanning, but the participant will wear proper ear protection. Some participants may experience claustrophobia during the scan. If the participant has steatosis on both MRS, he will be offered a referral to the Department of Gastroenterology.

Penetrations of skin (blood puncture and intravenous catheter insertion and insertion of sensor for continuous glucose monitoring) are associated with mild discomfort and risk of hematomas. A theoretical complication to skin penetration is superficial phlebitis. The condition is not dangerous and will be treated with antibiotics should any sign of infection be present. The risk of superficial phlebitis is small and minimized by following clinical standards for the insertion of intravascular catheters including double wiping of the involved skin with disinfectant alcohol and other sterile procedures.

The total blood loss will amount to approximately 365 ml distributed over a minimum of 2 weeks, which is not in any way harmful for the participant. Only participants with haemoglobin >7.5 mmol/l can participate, and all participants are offered iron treatment after the trial.

PARTICIPANTS PHYSICAL AND MENTAL INTEGRITY AND PRIVACY Information regarding participants of the project will be protected in accordance with the applicable laws of Denmark including the law concerning the processing of personal data. We will seek approval of the protocol by the Danish "Datatilsynet" via the The Capital Region of Denmark. The trial will follow the rules in European Union's General Data Protection Regulation.

The protocol complies with the Helsinki Declaration (Seventh revision 2013).

OPERATING COSTS AND ECONOMY The project is currently not supported by any medical companies and the responsible physician of the project has no economical affiliations with private companies, foundations or the like with interests in the research project. When funding for the project is in place the Research Ethics Committees will be notified.

AVAILABILITY OF DATA FOR PARTICIPANTS All participants are guaranteed access to more information about the project. Contact: Dr. Pernille Høgh Hellmann, MD, Center for Clinical Metabolic Research, Gentofte Hospital, DK-2900 Hellerup; e-mail: pernille.hoegh.hellmann@regionh.dk; Phone: +45 20911792.

ADJOURNMENT OF TRIAL Any participant can be withdrawn from the trial at any time, in case investigator finds it unsafe for the participant to continue. Also, the participant can be withdrawn if the participant meets any of the exclusion criteria, if compliance is insufficient (if participant has missed more than ¼ of planned doses, controlled at telephone call at day 5, 6 or 7 in the intervention period and at the end-of-intervention visit) evaluated by investigator, or in case exceptional circumstances make it impossible to complete the study. Likewise, any extraordinary event that makes it impossible to finish the project will result in termination of ongoing experiments. In all cases, the participant will be informed about the decision and the reason why. The participant may, at any time during the trial, voluntarily discontinue participation. In case of drop-outs, we will include new participants until we have 12 completers in each group.

THE RESEARCH GROUP Pernille Høgh Hellmann MD, Jonatan Ising Bagger PhD MD, Katrine Bagge Hansen PhD MD, Professor Tina Vilsbøll DMSc MD, Professor Filip Krag Knop PhD, MD

RECRUITMENT OF PARTICIPANTS Participants are recruited through the following methods: 1) Advertisement in newspapers or local newspapers or at www.forsøgsperson.dk. 2) Advertisement through flyers and posters. 3) Participants who participated in studies in the department in the past and gave consent that they would like to be contacted again in regard to participation in new studies in the department.

Participants who responded on advertisements will receive written information on e-mail or regular mail, whatever is preferred. All participants will also receive the leaflet "Forsøgspersonens rettigheder i et sundhedsvidenskabeligt forskningsprojekt" from the Ethical Committee in Denmark, august 2014.

After at least two days, the participant will be contacted by telephone and asked if he wants to participate in the study. If the participant has any questions, these will be answered as thoroughly as possible. If the participant is interested in participation, a time and place for the information visit will be scheduled. During the phone call, the participant is informed about the possibility to be accompanied by a person of own choice to all the visits during the trial.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) >24.9 kg/m2, If participant is included during COVID19-pandemic, maximum BMI is 32 kg/m2
* Haemoglobin ≥7.5 mmol/l
* Written informed consent

Exclusion Criteria:

If the participant is screened during COVID19, extra exclusion criteria is age>59 years.

If the participant is screened during COVID19-pandemic, following exclusion criteria is also applicable: 1) Diagnosed with asthma requiring medication or having uncontrolled asthma. 2) Beeing a current smoker. 3) diagnosed with hypertension. 4) having a job or engaging in daily activities, where it is not possible to adhere to the required distance of one meter to other people, judged by the investigator. 5) bA1c above 42 mmol/mol at screening.

* Use of glucose-lowering drugs, lipid-lowering drugs, warfarin, clopidogrel or non-vitamin K anti-coagulants
* Frequent use of anti-inflammatory drugs the last two months prior to inclusion, judged by the investigator
* Treatment with drugs with potential steatogenic side-effects within two months prior to inclusion
* Use of medication known to interact with prednisolone
* Use of curcumin-containing food supplements or other natural products that could cause confounding as evaluated by investigator
* Any regular drug treatment that cannot be discontinued for minimum 18 hours
* Previous diagnosis of T2D
* Diabetes (HbA1c ≥ 48 mmol/mol) found at screening
* Known viral, inherited or alcoholic liver disease, or any other condition known to affect liver
* Intake of more than 21 units of alcohol per week
* Nephropathy (eGFR < 60 ml/min/1.73 m² and/or urine albumin > 20 mg/l)
* In a weight management program, or planning to change life style, alcohol habits or eating habits during the course of the study
* Implanted metal objects contraindicative of MRS Claustrophobia
* Any condition that the investigator think would interfere with trial participation or with the safety of the participant.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only males are included
Enrollment: 24 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-06-07 (Actual); Study Completion 2021-06-11 (Actual)

PRIMARY OUTCOMES:
HOMA-IR | 12-14 days
  homeostatic model assessment of insulin resistance is calculated before and after intervention

SECONDARY OUTCOMES:
steatosis | 12-20 days
  Measured by MR spectroscopy of the liver (unit: %)
liver stiffness | 12-14 days
  Measured by FibroScan (unit: kPa)
concentration of alanine transaminase | 12-14 days
  Blood sample
concentration of aspartate transaminase | 12-14 days
  Blood sample
concentration of creatine kinase | 12-14 days
  Blood sample
glucagon levels under oral glucose tolerance test | 12-14 days
  Blood sample
concentration of amino acids under oral glucose tolerance test | 12-14 days
  Blood sample
urea concentration in plasma | 12-14 days
  Blood sample
urea concentration in urin | 12-14 days
  Urin sample
urea production | 12-14 days
  Estimated by collecting urin for 4-5 hours, measuring volume of urine and urea concentration
concentration of gamma glutamyl transferase | 12-14 days
  Blood sample
concentration of blood lipids | 12-14 days
  Blood sample
gut hormone concentration during oral glucose tolerance test | 12-14 days
  blood sample
concentration of inflammation markers (interleukines and high sensitivity CRP and TNF alpha) | 12-14 days
  blood sample
concentration of serum biomarkers of non-alcoholic steatohepatitis | 12-14 days
  blood sample
concentration of serum biomarkers of fibrosis in the liver | 12-14 days
  blood sample
concentration of fasting glucose | 12-14 days
  blood sample
concentration of glucose levels during oral glucose tolerance test | 12-14 days
  blood sample
concentration of serum bone markers | 12-14 days
  blood sample
concentration of fibroblast growth factors | 12-14 days
  blood sample
Gut microbiota analysis (abundance) | 12-20 days
  Feces sample before and after intervention
Gut microbiota analysis (alpha and beta diversity) | 12-20 days
  Feces sample before and after intervention
Gut microbiota analysis (link to phenotype of interest) | 12-20 days
  Feces sample before and after intervention
Glucose measurement by continuous monitor | 11-14 days
  subcutaneously, interstitial measurement (concentration of glucose) every 15 minutes in the intervention period
intra ocular eye pressure in both eyes | 12-14 days
  icare 100 tonometer measurement (unit: mmHg)
BOdy composition (fat, water, skeletal muscle mass, fat-free mass) | 12-14 days
  measured by bioimpedance (units: kg and %)
visceral fat tissue amount | 12-20 days
  MR-spectroscopy measurement (unit: cm3 at L3-level, 1 cm thick slice)
subcutaneous fat tissue amount | 12-20 days
  MR-spectroscopy measurement (unit: cm3 at L3-level, 1 cm thick slice)
Body weight | 12-14 days
  Body weight (unit: kg)
Body mass index | 12-14 days
  (kg/m2)
waist circumference | 12-14 days
  (unit: cm)
hip circumference | 12-14 days
  (unit: cm)
Questionnaire during oral glucose tolerance test every 30 minutes and ten minutes after ad libitum meal: How hungry do you feel? Range: I'm not hungry at all - I've never been more hungry | 12-14 days
  visual analogue scale evaluation (no visible numbers/points, just a clear line)
Questionnaire during oral glucose tolerance test every 30 minutes and ten minutes after ad libitum meal: How full do you feel? Range: I have a big hole in my stomach - I can not eat one single bite more | 12-14 days
  visual analogue scale evaluation (no visible numbers/points, just a clear line)
Questionnaire during oral glucose tolerance test every 30 minutes and ten minutes after ad libitum meal: How filled up do you feel? Range: Not filled up at all - totally filled up | 12-14 days
  visual analogue scale evaluation (no visible numbers/points, just a clear line)
Questionnaire during oral glucose tolerance test every 30 minutes and ten minutes after ad libitum meal: How much do you think you can eat? Range: nothing at all - really much | 12-14 days
  visual analogue scale evaluation (no visible numbers/points, just a clear line)
Questionnaire during oral glucose tolerance test every 30 minutes and ten minutes after ad libitum meal: How do you feel? Range: Really bad - really good | 12-14 days
  visual analogue scale evaluation (no visible numbers/points, just a clear line)
Questionnaire during oral glucose tolerance test every 30 minutes and ten minutes after ad libitum meal: do you feel nausious? Range: yes, very much - no, not at all | 12-14 days
  visual analogue scale evaluation (no visible numbers/points, just a clear line)
Questionnaire during oral glucose tolerance test every 30 minutes and ten minutes after ad libitum meal: How thirsty do you feel? Range: Not thirsty at all - very thirsty | 12-14 days
  visual analogue scale evaluation (no visible numbers/points, just a clear line)
Questionnaire during ad libitum meal: appearance of the meal: Range: Not appetizing - very appetizing | 12-14 days
  visual analogue scale evaluation (no visible numbers/points, just a clear line)
Questionnaire during ad libitum meal: Smell of the meal: Range: Not appetizing - very appetizing | 12-14 days
  visual analogue scale evaluation (no visible numbers/points, just a clear line)
Questionnaire during ad libitum meal: Taste of the meal: Range: Bad - Good | 12-14 days
  visual analogue scale evaluation (no visible numbers/points, just a clear line)
Questionnaire during ad libitum meal: Does the meal have unwanted taste? Range: no, not at all - yes, a lot | 12-14 days
  visual analogue scale evaluation (no visible numbers/points, just a clear line)
Questionnaire during ad libitum meal: How is the overall impression of the meal? Range: not appetizing - Very appetizing | 12-14 days
  visual analogue scale evaluation (no visible numbers/points, just a clear line)
Food consumption | 12-14 days
  Evaluated by calculating ingested meal at ad libitum meal at test days (unit: grams and calories)
systolic blood pressure | 12-14 days
  unit: mmHg
diastolic blood pressure | 12-14 days
  unit: mmHg
heart rate | 12-14 days
  Unit: beats per minute
resting energy expenditure (kcal/day) measured by inderect calorimetry | 12-14 days
  Measured for 15 minutes at test days.
Evaluation of food consumption the day before test day. Participant will fill out diary of all foods and drinks consumed. | 12-14 days
  24 hour recall questionnaire
Questionnaire regarding fullness before bedtime the day before test day: how hungry were you before bed time? Range: Very hungry - not hungry at all | 12-14 days
  Visual analogue scale (no points/number visible, just a clear line)
Evaluation of physical activity the day before test day. Participant will fill out diary of all physical activities including activity intensity. | 12-14 days
  24 hour recall questionnaire
concentration of c-peptide during oral glucose tolerance test | 12-14 days
  blood sample
concentration of lactate dehydrogenase | 12-14 days
  blood sample
concentration of free fatty acids during oral glucose tolerance test | 12-14 days
  blood sample
concentration of alkaline phosphatase | 12-14 days
  blood sample
concentration of albumin | 12-14 days
  blood sample
concentration of insulin fasting | 12-14 days
  blood sample
levels of insulin during oral glucose tolerance test | 12-14 days
  blood sample
thromboelastography measurement. | 12-14 days
  Blood sample
concentration of von Willebrands Factor in plasma | 12-14 days
  blood sample
concentration of protein C in plasma | 12-14 days
  blood sample
concentration of protrombin in plasma | 12-14 days
  blood sample
concentration of X-fib in plasma | 12-14 days
  Blood sample
concentration of PRO-C6 in plasma | 12-14 days
  blood sample
concentration of d-dimer in plasma | 12-14 days
  blood sample
concentration of fibrinogen in plasma | 12-14 days
  Blood sample

CONTACTS AND LOCATIONS:
Overall Officials: Filip K Knop, Professor, Principal Investigator — Gentofte university hospital, Hellerup, Denmark
Locations (1):
- Center for Clinical Metabolic Research, Hellerup, Denmark